CLINICAL TRIAL: NCT03997877
Title: Randomized Clinical Trial on the Effect of an Aerobic Exercise Program in Patients With Moderate-severe Sleep Apnea
Brief Title: Effect of an Aerobic Exercise Program in Patients With Moderate-severe Sleep Apnea
Acronym: SAH-2014
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAH-2014
Record Dates: First submitted 2019-06-19; First posted 2019-06-25 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Sleep Apnea Hypopnea Syndrome; Physical Activity
Keywords: sleep apnea syndrome; physical activity; mediterranean diet; metabolism; impact on sleep
MeSH Terms: conditions — Sleep Apnea, Obstructive; Motor Activity; Sleep Apnea Syndromes | interventions — Exercise; Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The usual physical activity valued by the YPAS questionnaire (Yale Physical Activity Survey) will be maintained. The questionnaire allows to calculate the time in physical activity expressed in hours / week, the energy expenditure expressed in MET-h / week and the summary index of physical activity that takes into account the frequency and duration of physical activity and oscillates from 0 to 137. A value below 51 identifies sedentary patients. Daily physical activity is controlled through a pedometer that measures the distance traveled daily by the patient and recorded in a walking book.
  The therapeutic control will be carried out by telephone call at the second and fourth month of treatment and a face-to-face clinical control at 3 and 6 months.
  Interventions: Other: Physical activity
- Intervention (Experimental): It is intended that the exercise program have a duration of 6 months and its realization does not suppose an excessive consumption of resources. Therefore, it must have a series of characteristics: low supervision and easily realizable by all patients, which implies flexibility in the schedule and without the need for instruments or special facilities. In this sense the walk is adjusted to these assumptions and the goal of 10.000 steps / day can encourage compliance.
  The subjects assigned to the intervention group will be supervised and trained by a physiotherapist who will explain the training program and resolve the doubts raised by the patient.
  Daily physical activity is controlled through a pedometer that measures the distance traveled daily by the patient and recorded in a walking book.
  The therapeutic control will be carried out by telephone call at the second and fourth month of treatment and a face-to-face clinical control at 3 and 6 months.
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — Increase physical activity Balanced diet
  Other Names: Mediterranean diet

SUMMARY:
In this paper, it is postulated that in sedentary patients with moderate-severe sleep apnea diagnosed by a sleep test, an increase in physical activity stimulated by the use of a pedometer during a period of 6 months can reduce the severity of OSAS by decreasing the number of respiratory events during sleep and when controlling for vascular risk factors.

DETAILED DESCRIPTION:
It is postulated that in sedentary patients with moderate to severe sleep apnea, an increase in physical activity can reduce the severity of OSAS.

Our main objective was to determine the effectiveness of a physical exercise program to reduce the number of respiratory disorders during sleep (AHI) in patients with moderate-severe OSAS. The primary outcome variable will be the decrease in the AHI at least 50% of its baseline value.

Secondary objectives were:

1. To evaluate the impact of a physical activity program on glucose metabolism (glycemia, insulinemia, glycosylated hemoglobin, HOMA index).
2. Determine the effect of the physical activity program on the lipid profile (total cholesterol, HDL-C, LDL-C, triglycerides, apolipoproteins A1 and B).
3. Assess the role of a physical activity program on the systolic and diastolic blood pressure.
4. Determine the effect of a physical activity program on body weight (BMI).
5. To analyze the effect of a physical activity program on the perception of the impact of sleep on daily life (FOSQ questionnaire).

It is a controlled, randomized and parallel group clinical trial with an allocation ratio of 1: 1 For randomization, a table of random numbers with sampling module of the Epidat 3.1 program will be prepared by a statistician who does not participate in the study.

The ratio of subjects assigned to each group will be 1: 1. The random numbers will be kept in closed envelopes.

The staff of the Sleep Unit will be responsible for explaining the result of the polygraphy and following the patient, but in no case will participate in the measurement of the results.

All patients will be informed about the nature of the clinical trial, but without exposing the hypothesis to the patient. There will be no differences in the patient's follow-up because it will be performed by the same physician.

Special emphasis will be made so that the medical and nursing staff does not try to obtain or offer specific information that may indicate to which treatment arm the patient was assigned.

Once the patient is randomized and assigned to an arm of the study, those assigned to the intervention group will be sent to the physiotherapist to explain and initiate the exercise program while the control group will be informed to maintain their usual physical activity.

All subjects will be recommended to maintain a stable sleep habit, to sleep at least 7 hours at night, avoid the intake of relaxing medication during the evening and maintain the nutritional pattern recommended by the American Heart Association, this is 35% of calories in the form of fat (22% monounsaturated fat, 6% polyunsaturated fat, 7% saturated fat) 15% proteins and 50% carbohydrates. These recommendations and an explanatory leaflet based on the pyramid model of the mediterranean diet will be delivered to the two groups. The monitoring of the diet will be supervised by filling in the questionnaire of the Quality Index of the Mediterranean Diet (KIDMED) by the subjects in the initial visit, the third month and the sixth month. In the initial visit, the type of diet will be evaluated and all patients will be advised to follow a mediterranean diet as a general treatment measure. If the Kidmed index is ≤ 3, it will be re-educated to perform a Mediterranean diet and if the index is ≥ 7 you will be advised to maintain the diet during the following months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Low physical activity (total duration <60 minutes / week or a physical activity index calculated using the YPAS scale <51).
* An AHI> 15 and <30 / hour or AHI> 30 and rejection of CPAP.
* Signature of the informed consent form.

Exclusion Criteria:

- Suspicion or knowledge of a chronic disease that prevents a physical exercise program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Change of the variable AHI measured by polygraphy | six months
  Decrease in the value of the AHI after a physical exercise program

SECONDARY OUTCOMES:
Changes in glucose metabolism after a physical exercise program. | six months
  Decrease in the value of glycemia, insulinemia, glycosylated hemoglobin and HOMA index
Changes on the lipid profile after a physical activity program | six months
  Decrease in the value of total cholesterol, HDL-C, LDL, triglycerides, apolipoprotein A-1 and B
Change in systolic and diastolic blood pressure values after a physical activity program. | six months
  The value of the blood pressure will be an average value of three blood pressure determinations
Change on body weight after a physical activity program | six months
  Value of the body mass index
Modification of daytime sleepiness after a physical activity program. | six months
  Change in daytime sleepiness measured by the Epworth Sleepiness Scale. The Epworth Scale includes 8 questions about the possibility of falling asleep in various situations, such as reading, watching television, talking, driving. Each question has four possible answers, with values between 0 and 3. The total score is obtained by adding the values of each answer option; the minimum value is zero (no sleepiness) and the maximum is 24, which means excessive sleepiness.
Change in the impact of sleep on daily living after a physical activity program | six months
  Change in the impact of daytime sleepiness on activities of daily living after a physical activity program by the Functional Outcomes of Sleep Questionnaire. The FOSQ consists of 30 questions divided into 5 subscales: general productivity, social activity, activity level, surveillance and sexual relations and intimacy. Each element has 4 possible answers: "without difficulty", "small difficulty", "moderate difficulty" and "a lot of difficulty". In some items, there is an alternative response if that the activity is not performed for other reasons unrelated to sleepiness. The scores of each one of the dimensions are obtained by means of the average of the items that form it. Items that have not been answered are not included. The score of each dimension has a minimum value of 0 (maximum functional impact) and a maximum value of 24 (no impact). The general score is obtained by adding the scores of each of the 5 dimensions and has a value between 0 and 120.

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Feu, MD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
The individual data will be available after deidenttification (text, tables, figures and appendices) to those researchers who provide a methodologically sound proposal and for meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available after the end of the study until one year the article publication.
Access Criteria: To obtain the data, a proposal must be sent to uicec@imibic.org. To gain access, data requestors will need to sign a data access agreement.